CLINICAL TRIAL: NCT07010965
Title: SAVE-PCI is a Prospective, Multi-center, Randomized Controlled Trial Evaluating the Safety and Efficacy of NyokAssist™ , a Small-bore Percutaneous Ventricular Assist Device (pVAD), in Comparison With Intra-aortic Balloon Pump (IABP) in Patients Undergoing Elective High-risk Percutaneous Coronary Intervention (PCI)
Brief Title: SAVE-PCI: NyokAssist™ Small-Bore VAD vs. IABP in Elective High-Risk PCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: magAssist, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-133(2)
Record Dates: First submitted 2025-05-28; First posted 2025-06-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-06

CONDITIONS: High-Risk PCI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NyokAssist™ (Experimental)
  Interventions: Device: NyokAssist™
- IABP Intra-aortic balloon pump (Active Comparator)
  Interventions: Device: IABP Intra-aortic balloon pump

INTERVENTIONS:
Device: NyokAssist™ — The NyokAssist™ Ventricular Assist Device can be placed across the aortic valve using a single femoral site. The device pumps blood from the left ventricle into the ascending aorta .
  Arms: NyokAssist™
Device: IABP Intra-aortic balloon pump — IABP uses counterpulsation to provide coronary flow
  Arms: IABP Intra-aortic balloon pump

SUMMARY:
SAVE-PCI is a prospective, multi-center, randomized controlled trial evaluating the safety and efficacy of NyokAssist™, a small-bore percutaneous ventricular assist device (pVAD), in comparison with intra-aortic balloon pump (IABP) in patients undergoing elective high-risk percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

1. Age eligible (18 ≤ Age ≤ 80)
2. Subject is indicated for a non-emergent percutaneous treatment of at least one de novo or restenotic lesion in a native coronary vessel or bypass graft .
3. Patient presence at least one of the following a or b:

   1. Intervention on an unprotected left main coronary artery or intervention on the last patent coronary artery .
   2. Intervention on patient presenting with three-vessel* disease.

      * Three-vessel disease was defined as the presence at least one sign ficant stenosis ≥ 50% in the left anterior descending artery (LAD) and/or side branch, left circumflex artery (LCX) and/or side branch, and right coronary artery (RCA) and/or side branch. In the case of left coronary artery dominance, a lesion ≥ 50% in the proximal LAD and the LCX qualified as three-vessel disease.
4. Ejection Fraction ≤40% or Coronary rotational atherectomy or According to the assessment of the cardiac team, PCI requires hemodynamic support .
5. Volunteered to participate and Signed Informed Consent and able to cooperate with the whole trial process.

Exclusion Criteria:

1. Acute ST elevation Myocardial Infarction within 24 hours or CK-MB that have not normalized after acute ST elevation Myocardial Infarction.
2. Pre-procedure cardiac arrest within 24 hours of enrollment requiring CPR.
3. Subject is in cardiogenic shock defined as:

   * CI < 2.2 L/min/m2 and PCWP > 15 mmH
   * Hypotension (systolic BP < 90 mmHg for >30 minutes or the need for supportive measures to maintain a systolic BP of greater than or equal to 90 mmHg) AND end organ hypoperfusion (cool extremities OR [a urine output of < 30 mL/hour AND a HR > 60 BPM])
4. Mural thrombus in the left ventricle.
5. The presence of aortic valve replacement or mechanical circulatory support device.
6. Subject has mechanical complications of myocardial infarction.
7. Documented presence of severe aortic stenosis.
8. Documented presence of moderate to severe mitral stenosis.
9. Documented presence of severe aortic insufficiency.
10. Severe peripheral arterial obstructive disease that would preclude device placement.
11. Abnormalities of the aorta that would preclude surgery, including aortic aneurysms,aortic dissection and extreme tortuosity or calcifications.
12. Subject with renal failure (creatinine ≥265μmol/L)
13. Subject with liver dysfunction ( liver enzymes and bilirubin levels ≥3x ULN )
14. Subject has uncorrectable abnormal coagulation parameters (platelet count ≤ 75╳109 /L or fibrinogen ≤ 1.50 g/L)
15. History of recent (within 1 month) stroke or TIA .
16. Severe right ventricular dysfunction,such as severe pulmonary hypertension.
17. Allergy or intolerance to heparin, aspirin, ADP receptor inhibitors or contrast media.
18. Subject with documented heparin induced thrombocytopenia.
19. Subject has pregnant or lactating.
20. Participation in the active follow-up phase of another clinical study of an investigational drug or device within 1 month.
21. Investigators consider unsuitable to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
MACCE-free rate | Device Delivery through 30 Days
  The Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) Free Rate

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Beijing Anzhen Hospital Capital Medical University, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Guangdong Provincial People's Hospital, Guangzhou
  - Nanfang Hospital Southern Medical University, Guangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - The First Hospital of Lanzhou University, Lanzhou
  - ZhongShan Hospital Fudan University, Shanghai
  - Peking University First Hospital Taiyuan Hospital, Taiyuan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen
  - Fuwai Yunnan Hospital Chinese Academy of Medical Science, Yunnan